CLINICAL TRIAL: NCT05015894
Title: Investigation of the Pharmacokinetics of Subcutaneously Administered NNC0480-0389 in Participants With Various Degrees of Impaired Renal Function Compared to Participants With Normal Renal Function
Brief Title: A Research Study Looking Into Blood Levels of the Medicine NNC0480-0389 in Participants With Reduced Kidney Function Compared to Participants With Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9389-4682; 2021-001450-57 (EudraCT Number); U1111-1266-0594 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-08-19; First posted 2021-08-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NNC0480-0389 (Experimental): All participants will be administered a single s.c. dose of 18 mg NNC0480-0389
  Interventions: Drug: NNC0480-0389

INTERVENTIONS:
Drug: NNC0480-0389 — A single dose of 18 mg NNC0480 0389 administered subcutaneously (under the skin).
  Total duration of study participation for each participant is 38 to 66 days

SUMMARY:
Novo Nordisk is developing a combination therapy with the study medicine NNC0480-0389 and an already approved medicine called "semaglutide" for the treatment of type-2 diabetes (T2D). It is expected that the combination will further improve the blood sugar control compared to semaglutide therapy alone.In this study the blood levels of NNC0480-0389 will be compared in people with various degrees of reduced kidney function to the blood levels in people with normal kidney function, after administration of one dose of 18 mg NNC0480-0389. Participants will only get the study medicine as two injections into a skinfold of participants belly (subcutaneous).

The study will last for about 65 days including a screening phase of up to 28 days prior to dosing.

If participants are eligible for the study, participants will have 11 visits to the study centre including one in-house stay of 5 days and 4 nights (Visit 2) and nine ambulatory visits (Visit 3 to Visit 11).

Participants' vital signs (heart rate, blood pressure, body temperature) will be measured, participants will have blood drawn, urine will be collected and electrocardiograms (ECGs) will be recorded.If participants are women and can get pregnant they cannot take part in the study. A hormone test will be done to check if participants may be post-menopausal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential, aged 18-75 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 20.0 and 39.9 kg/m^2 (both inclusive)
* Meeting the pre-defined GFR criteria using estimated GFR (eGFR) based on serum creatinine for any of the renal function groups:

  * For participants with normal renal function: eGFR of equal to or greater than 90 mL/min
  * For participants with mild renal impairment: eGFR of 60-89 mL/min
  * For participants with moderate renal impairment: eGFR of 30-59 mL/min
  * For participants with severe renal impairment: eGFR of 15-29 mL/min not requiring dialysis
  * For participants with kidney failure: eGFR of less than 15 mL/min or requiring dialysis treatment

Specific inclusion criteria for participants with kidney failure requiring dialysis treatment:

* Current treatment with haemodialysis

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs, or non-routine vitamins, which at the investigators judgement may affect participant safety or the results of the study within 14 days before screening.
* Use of drugs known to affect creatinine clearance including cephalosporin and aminoglycoside antibiotics, flucytosine, cisplatin, cimetidine, trimethoprim and cibenzoline within 14 days or 5 half-lives, whichever is greater, before dosing the investigational medicinal product (IMP).
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions (except conditions associated with renal impairment or kidney failure).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
AUC0-∞,NNC0480-0389,SD, area under the NNC0480-0389 plasma concentration time curve after a single dose | From baseline (visit 2, day 1, pre-dose) until completion of the end-of-study visit (visit 11, day 36)
  h*nmol/L

SECONDARY OUTCOMES:
Cmax,NNC0480-0389,SD, Maximum observed NNC0480-0389 plasma concentration after a single dose | From baseline (visit 2, day 1, pre-dose) until completion of the end-of-study visit (visit 11, day 36)
  nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com